CLINICAL TRIAL: NCT00248170
Title: Comparison Trial of Letrozole to Anastrozole in the Adjuvant Treatment of Postmenopausal Women With Hormone Receptor and Node Positive Breast Cancer
Acronym: FACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345D2411; 2005-004263-35 (EudraCT Number); EUDRACT number 2005-004263-35 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; letrozole; anastrozole; adjuvant; postmenopausal; FACE
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole

ARMS (2):
- Letrozole (Experimental): 2.5 mg by mouth (p.o.) once daily
  Interventions: Drug: Letrozole
- Anastrozole (Active Comparator): 1 mg p.o. once daily
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Letrozole — 2.5 mg tablets
  Arms: Letrozole
Drug: Anastrozole — 1 mg tablets
  Arms: Anastrozole

SUMMARY:
Eligible patients will be post-menopausal hormone receptor- and lymph node-positive females who recently underwent primary surgery for breast cancer. Patients will be randomized to letrozole (2.5 mg per day for 5 years) vs anastrozole (1 mg per day for 5 years). Follow up will occur for 5 years after the completion of enrollment for survival and disease status updates.

ELIGIBILITY:
Inclusion Criteria:

* Recent primary surgery for breast cancer
* Early stage breast cancer
* Postmenopausal
* Hormone receptor positive
* Positive lymph node involvement

Exclusion Criteria:

* Metastatic disease
* Presence of contralateral breast cancer including DCIS
* Progression

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 33 Years to 96 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4172 (Actual)
Dates: Start 2005-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (239):
- United States (42):
  - Birmingham Hematology and Oncology Associates, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Northern Arizona Hematology/Oncology Associates, P.C., Flagstaff, Arizona
  - Oncology & Hematology Associates, PC, New London, Connecticut
  - Florida Cancer Specialists, Fort Meyers, Florida
  - Sarah Cannon Research Institute, Jacksonville, Florida
  - Cancer Centers of Florida PA, Ocoee, Florida
  - Florida Cancer Institute, Orlando, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Kansas City Cancer Center, Overland Park, Kansas
  - Wichita Community Clinical Oncology Program, Wichita, Kansas
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - St. Louis Cancer & Breast Institute, St Louis, Missouri
  - New York Oncology Hematology, P.C. NYOH Latham, Troy, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Aultman Cancer Center, Canton, Ohio
  - Sarah Cannon Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Oncology Associates of Oregon, PC, Eugene, Oregon
  - Medical Oncology Associates of Wyorning Valley, PC, Kingston, Pennsylvania
  - Chattanooga Oncology and Hematology Assoicates, PC, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - Texas Cancer Center ( Medical City Dallas Hospital), Dallas, Texas
  - Texas Oncology Presbyterian Hospital, Dallas, Texas
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Texas Oncology Texas Oncology PA, Dallas, Texas
  - Texas Cancer Center Denton, Denton, Texas
  - El Paso Cancer Treatment Ctr-East, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - San Antonio Tumor and Blood Clinic, Fredericksburg, Texas
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center- McAllen, McAllen, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Cancer Center- Sherman, Sherman, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer and Research Center, Waco, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Cancer Specialists, P.C., Vancover, Washington
- Australia (23):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Port Macquarie, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Tweed Heads, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Nambour, Queensland
  - Novartis Investigative Site, Redcliff, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Toorak Gardens, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, East Bentleigh, Victoria
  - Novartis Investigative Site, Epping, Victoria
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Franston, Victoria
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Dunedin
  - Novartis Investigative Site, Hamilton
- Austria (14):
  - Novartis Investigative Site, Graz, Austria
  - Novartis Investigative Site, Vienna, Austria
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Friesach
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Güssing
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Villach
  - Novartis Investigative Site, Wiener Neustadt
- Belgium (12):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Libramont
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Wilrijk
- Canada (7):
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- China (4):
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Denmark (10):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Herning
  - Novartis Investigative Site, Hillerød
  - Novartis Investigative Site, Næstved
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- France (14):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montbéliard
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Périgueux Cédex
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (26):
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, Amberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Witten
- Ireland (5):
  - Novartis Investigative Site, Galway, Ireland
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Letterkenny
  - Novartis Investigative Site, Limerick
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Litwinsky
- Italy (17):
  - Novartis Investigative Site, Montevarchi, AR
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Biella, BI
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Antella - Bagno A Ripoli, FI
  - Novartis Investigative Site, Forlì, FO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Castelfranco Veneto, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Fermo
- Japan (19):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Netherlands (5):
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Veldhoven
- Novartis Investigative Site, Skien, Norway
- South Korea (3):
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (9):
  - Novartis Investigative Site, Alicante, Alicante
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Zaragoza, Zaragoza
- Sweden (3):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Schaffhausen
  - Novartis Investigative Site, Winterthur
- United Kingdom (17):
  - Novartis Investigative Site, Hull, East Yorkshire
  - Novartis Investigative Site, Glasgow, Glasgow
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Chelmsford
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Merseyside
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Rhyl
  - Novartis Investigative Site, Sheffiled
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants, who had recently undergone surgery, were randomly assigned in 1:1 ratio to letrozole or anastrozole. Participants received daily treatment until disease recurrence/relapse or for a maximum of 5 years. Participants underwent post-treatment long term follow-up for disease-free survival and overall survival.
Period: Overall Study
Arm/Group | Letrozole | Anastrozole
Started | 2078 | 2094
Intent-to-treat (ITT) | 2061 | 2075
Safety Set | 2049 | 2062
Completed | 1317 | 1286
Not Completed | 761 | 808
Not completed — Withdrawal by Subject | 71 | 79
Not completed — Protocol Violation | 35 | 30
Not completed — Lost to Follow-up | 28 | 35
Not completed — Disease progression | 196 | 216
Not completed — Death | 28 | 47
Not completed — Adverse Event | 311 | 296
Not completed — Administrative problems | 22 | 25
Not completed — Abnormal test procedure(s) result | 49 | 61
Not completed — Abnormal laboratory values | 4 | 0
Not completed — Protocol deviation | 17 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Anastrozole | Total
Number analyzed (Participants) | 2061 | 2075 | 4136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.48) | 63.1 (8.45) | 63.2 (8.46)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 2061 | 2075 | 4136

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: Disease-free survival was defined as the time from the date of randomization to the date of the first documentation of re-occurrence of invasive breast cancer in local, regional or distant sites, new invasive breast cancer in the contra-lateral breast, or death from any cause.
Time Frame: 84 months
Population: Intent-to-treat (ITT) - the ITT contained randomized participants who had no protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2061 | 2075
Months | NA [84.14 to NA] — The median was not reached and therefore, could not be calculated. | NA [NA to NA] — The median was not reached and therefore, could not be calculated.
Statistical Analysis 1: Comparison: Letrozole vs Anastrozole; Test type: Superiority or Other; p = 0.3150, Log Rank

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: 84 months
Population: Intent-to-treat (ITT) - the ITT contained randomized participants who had no protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2061 | 2075
Months | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated. | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated.

3. Secondary Outcome: Time to Development of Distant Metastases
Description: Time to development of distant metastases was defined as the time from date of randomization to the date of the first development of any recurrent or metastatic disease in sites other than the local mastectomy scar, the ipsilateral breast in case of breast conservation or the contra lateral breast.
Time Frame: 84 months
Population: Intent-to-treat (ITT) - the ITT contained randomized participants who had no protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2061 | 2075
Months | NA [84.14 to NA] — The median was not reached and therefore, the median could not be calculated. | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated.

4. Secondary Outcome: Time to Development of Contra Lateral Breast Cancer
Description: Time to development of contra lateral breast cancer was defined as the time from the date of randomization to the date of the first development of any disease in the contra lateral breast.
Time Frame: 84 months
Population: Intent-to-treat (ITT) - the ITT contained randomized participants who had no protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2061 | 2075
Months | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated. | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated.

5. Secondary Outcome: Distant Disease-free Survival
Description: Distant disease-free survival was defined as the time from date of randomization to the date of the first development of any relapse at a distant site or death from any cause.
Time Frame: 84 months
Population: Intent-to-treat (ITT) - the ITT contained randomized participants who had no protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2061 | 2075
Months | NA [84.14 to NA] — The median was not reached and therefore, the median could not be calculated. | NA [NA to NA] — The median was not reached and therefore, the median could not be calculated.

6. Secondary Outcome: Change From Baseline in Serum Lipid Profiles
Description: Total cholesterol was analyzed to assess the impact on serum lipids profiles. The adjusted means was calculated.
Time Frame: baseline, 6, 12, 24, 36, 48 and 60 months
Population: Safety Set: The safety set included randomized participants who received at least one of study medication and had at least one post baseline assessment.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2049 | 2062
mg/dL
  6 months | 5.643 [5.584 to 5.701] | 5.553 [5.495 to 5.611]
  12 months | 5.569 [5.510 to 5.629] | 5.511 [5.452 to 5.570]
  24 months | 5.508 [5.445 to 5.572] | 5.436 [5.373 to 5.499]
  36 months | 5.429 [5.359 to 5.500] | 5.427 [5.357 to 5.497]
  48 months | 5.395 [5.323 to 5.468] | 5.366 [5.293 to 5.438]
  60 months | 5.375 [5.300 to 5.451] | 5.368 [5.292 to 5.443]

7. Secondary Outcome: Percentage of Participants Who Experienced Clinical Fracture Events
Description: The incidence of clinical fractures was analyzed.
Time Frame: 84 months
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2049 | 2062
Percentage of participants | 9.3 | 8.1

8. Secondary Outcome: Percentage of Participants Who Experienced Cardiovascular Events
Description: The incidence of ischemic heart disease, cardiac failures, cerebrovascular accidents and thromboembolic events was analyzed.
Time Frame: 84 months
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 2049 | 2062
Percentage of participants
  Ischemic heart disease | 2.4 | 1.5
  Cardiac failures | 1.5 | 0.7
  Cerebrovascular accidents | 1.6 | 1.5
  Thromboembolic events | 1.2 | 1.2

ADVERSE EVENTS:
Groups:
- Letrozole: Letrozole
- Anastrozole: Anastrozole
Arm/Group | Letrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 486/2049 | 520/2062
Other Adverse Events (participants affected / at risk) | 1747/2049 | 1762/2062
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=2049) | Anastrozole (N=2062)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 4
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 8 | 8
Angina unstable (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 19 | 15
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Bundle branch block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 4
Cardiac disorder (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 9 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 9 | 4
Cardiac fibrillation (Cardiac disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 7 | 2
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Gastrocardiac syndrome (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 4
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Palpitations (Cardiac disorders) | 1 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Syndactyly (Congenital, familial and genetic disorders) | 0 | 1
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 8 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 2
Autoimmune thyroiditis (Endocrine disorders) | 2 | 0
Goitre (Endocrine disorders) | 4 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 9 | 2
Dacryostenosis acquired (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Lens dislocation (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 2 | 1
Open angle glaucoma (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 5
Abdominal pain lower (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Anal sphincter atony (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 5
Gastritis erosive (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 3 | 3
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 7 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 11 | 6
Oesophagitis (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Spigelian hernia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 2
Tooth loss (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 6
Asthenia (General disorders) | 0 | 6
Cardiac death (General disorders) | 2 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Death (General disorders) | 2 | 2
Device damage (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 2
Device malfunction (General disorders) | 0 | 1
Disease progression (General disorders) | 2 | 2
Disease recurrence (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Fat necrosis (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 4 | 3
Impaired healing (General disorders) | 1 | 1
Implant site extravasation (General disorders) | 1 | 0
Injection site phlebitis (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 3
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Patient-device incompatibility (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 8
Sudden death (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 7 | 5
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 8 | 11
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 5
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 0 | 2
Breast abscess (Infections and infestations) | 1 | 1
Breast cellulitis (Infections and infestations) | 6 | 4
Bronchitis (Infections and infestations) | 3 | 4
Bronchopneumonia (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 8 | 9
Clostridium difficile colitis (Infections and infestations) | 3 | 3
Cystitis (Infections and infestations) | 2 | 3
Device related infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 7
Encephalitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 5 | 8
Escherichia sepsis (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 7 | 2
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Incision site abscess (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 2 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Lymphangitis (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 2 | 5
Meningitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 2
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 16 | 29
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 2 | 2
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyometra (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 3 | 8
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 3
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 8
Urosepsis (Infections and infestations) | 3 | 3
Vaginal infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 3 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 14 | 10
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 17 | 13
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 8 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 3 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 5 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 9 | 6
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 4
Multiple fractures (Injury, poisoning and procedural complications) | 3 | 3
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 3
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 2
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Radiation pericarditis (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 2 | 7
Rib fracture (Injury, poisoning and procedural complications) | 3 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 4
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 0
Tracheal injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 5
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 6 | 3
Amylase increased (Investigations) | 0 | 1
Aspiration pleural cavity (Investigations) | 1 | 0
Biopsy breast (Investigations) | 0 | 2
Biopsy lymph gland (Investigations) | 1 | 0
Bone density decreased (Investigations) | 1 | 0
Carbohydrate antigen 15-3 increased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 2 | 1
Lipase increased (Investigations) | 0 | 1
Mammogram abnormal (Investigations) | 1 | 0
Mediastinal biopsy (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 6
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 15
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retro-orbital neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 6
Cerebral amyloid angiopathy (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 6
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 5
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 3
Dementia (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 6
Dysarthria (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 4
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Horner's syndrome (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypogeusia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 2
Sensory loss (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Spinal epidural haemorrhage (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 4
Syncope (Nervous system disorders) | 13 | 4
Tardive dyskinesia (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 8 | 5
Tremor (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 8
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 9 | 11
Drug dependence (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 3 | 2
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0
Somatisation disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 7
Renal failure acute (Renal and urinary disorders) | 6 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 4
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1
Anisomastia (Reproductive system and breast disorders) | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 1 | 0
Breast fibrosis (Reproductive system and breast disorders) | 0 | 2
Breast haematoma (Reproductive system and breast disorders) | 1 | 1
Breast inflammation (Reproductive system and breast disorders) | 0 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 2
Breast oedema (Reproductive system and breast disorders) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 1
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 5 | 3
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 2
Uterine fistula (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 2 | 1
Uterine prolapse (Reproductive system and breast disorders) | 2 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 1
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 1
Breast lump removal (Surgical and medical procedures) | 1 | 0
Breast operation (Surgical and medical procedures) | 1 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 5 | 10
Breast prosthesis removal (Surgical and medical procedures) | 1 | 1
Breast reconstruction (Surgical and medical procedures) | 24 | 16
Central venous catheter removal (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 6 | 3
Mastectomy (Surgical and medical procedures) | 5 | 6
Mechanical ventilation (Surgical and medical procedures) | 0 | 1
Medical device removal (Surgical and medical procedures) | 1 | 0
Meniscus removal (Surgical and medical procedures) | 1 | 0
Modified radical mastectomy (Surgical and medical procedures) | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0
Scar excision (Surgical and medical procedures) | 0 | 2
Spinal laminectomy (Surgical and medical procedures) | 0 | 1
Wound treatment (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 2 | 1
Aortic stenosis (Vascular disorders) | 2 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Capillary fragility (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 3 | 4
Deep vein thrombosis (Vascular disorders) | 2 | 8
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 2 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 4
Hypertensive crisis (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 3 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 2 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=2049) | Anastrozole (N=2062)
Nausea (Gastrointestinal disorders) | 127 | 148
Fatigue (General disorders) | 345 | 341
Oedema peripheral (General disorders) | 100 | 104
Radiation skin injury (Injury, poisoning and procedural complications) | 120 | 88
Hypercholesterolaemia (Metabolism and nutrition disorders) | 155 | 151
Arthralgia (Musculoskeletal and connective tissue disorders) | 983 | 983
Back pain (Musculoskeletal and connective tissue disorders) | 207 | 187
Bone pain (Musculoskeletal and connective tissue disorders) | 138 | 120
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 122 | 144
Myalgia (Musculoskeletal and connective tissue disorders) | 232 | 211
Osteopenia (Musculoskeletal and connective tissue disorders) | 202 | 172
Osteoporosis (Musculoskeletal and connective tissue disorders) | 221 | 224
Pain in extremity (Musculoskeletal and connective tissue disorders) | 167 | 174
Dizziness (Nervous system disorders) | 92 | 107
Headache (Nervous system disorders) | 127 | 164
Depression (Psychiatric disorders) | 141 | 129
Insomnia (Psychiatric disorders) | 160 | 149
Cough (Respiratory, thoracic and mediastinal disorders) | 106 | 120
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 111 | 92
Alopecia (Skin and subcutaneous tissue disorders) | 126 | 134
Hot flush (Vascular disorders) | 666 | 666
Hypertension (Vascular disorders) | 152 | 145
Lymphoedema (Vascular disorders) | 158 | 177

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.